CLINICAL TRIAL: NCT03389425
Title: Application of the Simplified Intervention to Modify Physical Activity, Lifestyle, and Eating Behavior From Dr. Cenk Tek and Colleagues of Yale University to a Sample of Obese Patients With Stable Schizophrenia or Schizoaffective Disorder on Antipsychotic Medications in the Pathways to Housing Multidisciplinary Care Setting: A Feasibility Study
Brief Title: Application of the SIMPLE Program for Weight Loss at Pathways to Housing: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB14-1546
Record Dates: First submitted 2017-12-21; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Abdominal Obesity
MeSH Terms: conditions — Obesity; Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIMPLE weightloss group (Experimental)
  Interventions: Behavioral: simplified intervention to modify physical activity, lifestyle, and eating behavior

INTERVENTIONS:
Behavioral: simplified intervention to modify physical activity, lifestyle, and eating behavior — 16 week, behavioural weightloss intervention.

SUMMARY:
The objective of this study is to assess feasibility of the application of an adapted version, with permission, of Dr. Cenk Tek's Simplified Intervention to Modify Physical activity, Lifestyle, and Eating behavior (SIMPLE Program), at Pathways to Housing in Calgary, Alberta.

Dr. Tek and his colleagues reviewed the literature and eloquently summarized how individuals with severe mental illness, particularly schizophrenia and schizoaffective disorder are disproportionately affected by obesity and its cardio-metabolic sequelae leading to markedly reduced longevity and increased healthcare costs. Most new antipsychotic medications, which are credited for significant advances in patients' quality of life, appear to induce further weight gain, compounding the problem of obesity and related medical morbidity and mortality. In addition to the weight gain associated with psychiatric medications, sedentary life style, lack of availability of healthy food options, poverty, low level of physical activity, cigarette smoking, and inadequate knowledge or understanding of health maintenance, appear to contribute to the increased obesity rates and poor health in the severely mentally ill.

Dr. Tek and colleagues reviewed the available literature on weight loss interventions in individuals with severe mental illness. Despite the overwhelming problems related to obesity, Dr. Tek's team found that research on obesity interventions for persons with schizophrenia is relatively neglected and that there were no treatments that were convincingly shown to be effective for weight reduction in this population with unique needs. Sensing a major societal gap, they decided to create their own weight loss intervention specifically for individuals with severe mental illness. Toward this aim, they collaborated with Dr. Kelly Brownell who created the Lifestyle, Exercise, Attitudes, Relationships, and Nutrition or LEARN Program. This multi-faceted program is designed to promote positive changes in motivation, attitude and deeply ingrained habits that will lead to long lasting weight loss. Brownell's LEARN program is a self-directed weight loss program that empowers the user to make lifestyle changes. Dr. Tek and his colleagues modified and built upon the program by creating the Simplified Intervention to Modify Physical activity, Lifestyle, and Eating behavior or SIMPLE program specifically for individuals with severe mental illness (http://www.simpleprogram.org/).

The SIMPLE program is a group weight loss intervention designed for obese patients with schizophrenia or schizoaffective disorder. Dr. Tek and his team piloted their modified weight loss program and published their findings in 2007. Their preliminary study yielded greater weight loss than any of the published randomized controlled trials for a chronic and stable schizophrenia sample, and was the only study to show continued weight loss after the intervention ended. These early results prompted a new larger randomized controlled trial with the largest sample studied to date, an extended period of follow-up, and more detailed testing of the effects of weight loss on schizophrenia symptoms, quality of life, and laboratory markers of obesity related illness risk over a period of up to 16 months. Preliminary results of this trial show significant, sustained weight loss.

The goal of this study presented for ethics review, is to apply Dr. Tek's 16-week intervention to a small group of patients at the Pathways to Housing program in Calgary, Alberta. The study coordinator will use Dr. Tek's published manuals, giving full acknowledgment to the authors, to create weekly supportive educational sessions for the group of patients. Three Pathways to Housing staff members, who regularly create education groups for Pathways to Housing patients during a weekly "lifestyle group", will sit in on each session. Weight (to calculate BMI) and waist circumference will be measured weekly. There will be no control group. The proposed feasibility study is designed to fit seamlessly within existing frameworks at Pathways to Housing.

Upon completion of the study, we will convene a debriefing session with both the participants and the three Pathways to Housing staff to learn whether patients found the intervention valuable, and whether staff members feel capable of implementing the program on their own going forward. If the program is found to be feasible, the materials created will be available for future use by the multidisciplinary team at Pathways to Housing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be between 18 and 65 years of age.
2. Have a BMI of 28 or greater
3. Meet DSM-IV criteria for schizophrenia or schizoaffective disorder
4. Be on a stable dose of antipsychotic medication for at least one month, with positive symptoms stability as judged by the patient's medical doctors

Exclusion Criteria:

1. A history of dementia or mental retardation
2. Not capable of giving informed consent for participation in this study
3. Ongoing pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2015-10-08 (Actual)

PRIMARY OUTCOMES:
Weight | Weekly for 16 weeks, corresponding with each scheduled intervention group
  In Kilograms
Waist Circumference | Weekly for 16 weeks, corresponding with each scheduled intervention group
  In centimeters from midway between the iliac crest and lower rib
BMI | Weekly for 16 weeks, corresponding with each scheduled intervention group
  kg/ m squared

CONTACTS AND LOCATIONS:
Overall Officials: Vera H Krejcik, MD, Study Director — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SIMPLE program manuals — http://www.simpleprogram.org/